CLINICAL TRIAL: NCT03799939
Title: Chimney Trial - Randomized, Controlled, Multi Center Trial of Parastomal Hernia Prevention
Brief Title: Chimney Trial of Parastomal Hernia Prevention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Elisa Mäkäräinen, Principal Investigator, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 305/2018
Record Dates: First submitted 2019-01-06; First posted 2019-01-10 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Parastomal Hernia; Rectal Adenocarcinoma; Abdominoperineal Resection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Chimney trial is a prospective randomized controlled multicenter trial.
Who Masked: Participant
Masking Description: Participants are unaware of the randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Polyvinylidene fluoride mesh used in this trial (Dynamesh IPST) is synthetic mesh with central tube to accommodate bowel tightly and designed to prevent and treat parastomal hernia.
  Interventions: Device: Intervention group
- Control group (No Intervention): Participants in control group are operated with no preventive mesh.

INTERVENTIONS:
Device: Intervention group — Polyvinylidene fluoride mesh (Dynamesh IPST) is used on intraperitoneal onlay position to prevent parastomal hernia.
  Arms: Intervention group

SUMMARY:
Chimney trial is designed to compare the effectiveness and safety of specifically designated polyvinylidene fluoride mesh (PVDF, Dynamesh IPST) to controls in a multi center, randomized setting.

DETAILED DESCRIPTION:
The European Hernia Society recommends the use of prophylactic mesh when permanent colostomy is made. The results of previous trials using keyhole technique are partially unsatisfactory. Specifically designed PVDF mesh used in this trial showed promising results in previous small trial.

Chimney trial is designed to compare the effectiveness and safety of mesh group to controls operated with no preventive mesh in parastomal hernia prevention after laparoscopic or robotic-assisted abdominoperineal resection or low Haartman's procedure for rectal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Rectal adenocarcinoma with curative intent laparoscopic or robotic assisted abdominoperineal resection or low Hartmann´s operation and permanent colostomy
* Patient has a life expectancy of at least 12 months.
* Patient must sign Informed consent before any study procedures and agrees to attend all study visits

Exclusion Criteria:

* Abdominoperineal resection or Hartmann's operation by laparotomy or conversion to laparotomy
* Complication requiring laparotomy during post surgery treatment at surgical ward after APR
* Patient with a comorbid illness or condition that would preclude the use of surgery (ASA 4-5).
* Patients with concurrent or previous malignant tumors within 5 years before study enrollment
* Patients with T4b tumors which impose a multi-organ resection
* Rectal malignancy other than adenocarcinoma
* Patient undergoing emergency procedures
* Planned rectal surgery along with major concomitant procedures (e.g. hepatectomies, other intestinal resections).
* Metastatic disease with no possibility of curative surgery
* Pregnant or suspected pregnancy
* Patients living geographically distant and/or unwilling to return for follow-ups or comply with all study requirements
* Active abdominal infection at the time of surgery
* Previous surgery at the colostomy site
* Language barrier or other reasons why informed consent is not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of parastomal hernia | 12 months
  Incidence of parastomal hernia at 12 months follow up

SECONDARY OUTCOMES:
Incidence of parastomal hernia at long term follow up | 5 years
  Incidence of parastomal hernia during 5 years of follow up
Surgical site infection rate | 30 days
  Surgical site infections measured by Clavien-Dindo Classification
Complications | 30 days
  Complications measured by Clavien-Dindo Classification
Stoma related complications | 5 years
  Stoma related complications measured by Clavien-Dindo Classification
Reoperation rate | 5 years
  Need for reoperations
Operative time | 1 day
  Operative time
Length of stay | 30 days
  Length of stay at the hospital
Rand 36 quality of life | 5 years
  Quality of life measured by Rand-36 quality of life questionnaire
Quality of life measured by Colostomy impact score | 5 years
  Quality of life measured by Colostomy impact score
Medico-economic substudy | 5 years
  Medico-economic substudy including both short and long term costs included in both groups
Radiological substudy of stoma distance | 3 years
  Distance of stoma from midline defined by umbilicus
Radiological substudy of adipose tissue thickness | 3 years
  Thickness of adipose tissue on computer tomography scan on contralateral site of stoma

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Mäkäräinen-Uhlbäck, M.D., Principal Investigator — Oulu University Hospital
Locations (7):
- Finland (6):
  - Helsinki University Hospital, Helsinki
  - Keski-Suomi Central Hospital, Jyväskylä
  - Oulu University Hospital, Oulu
  - Seinäjoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Maziar Nikberg, Västerås, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Makarainen E, Wiik H, Nikberg M, Kossi J, Carpelan-Holmstrom M, Pinta T, Lehto K, Nikki M, Jarvinen J, Ohtonen P, Rautio T. Parastomal Hernia Prevention Using Funnel-Shaped Intra-Abdominal Mesh Compared to No Mesh: The Chimney Randomized Clinical Trial. JAMA Surg. 2024 Nov 1;159(11):1244-1250. doi: 10.1001/jamasurg.2024.3260. PMID 39196580
- [Derived] Makarainen-Uhlback E, Wiik H, Kossi J, Nikberg M, Ohtonen P, Rautio T. Chimney Trial: study protocol for a randomized controlled trial. Trials. 2019 Nov 28;20(1):652. doi: 10.1186/s13063-019-3764-y. PMID 31779699